CLINICAL TRIAL: NCT01516645
Title: Phase 1, Open-Label, Dose Escalation Study of Anti-CD98 Monoclonal Antibody KHK2898 as Monotherapy in Subjects With Advanced Solid Tumors Who No Longer Respond to Standard Therapy or For Whom No Standard Therapy Is Available
Brief Title: Phase 1 Study of KHK2898 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHK2898-001
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Solid Tumour
Keywords: Squamous cell type tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KHK2898 (Experimental)
  Interventions: Drug: KHK2898

INTERVENTIONS:
Drug: KHK2898 — injection

SUMMARY:
This is a two-part, Phase 1 open label, single-center, dose escalation study of KHK2898 as monotherapy in subjects with advanced solid tumors who no longer respond to standard therapy or for whom no standard therapy is available.

DETAILED DESCRIPTION:
The study will be conducted in two parts. In Part 1, a standard 3+3 designed dose escalation phase, subjects will receive KHK2898, administered intravenously, once every 2 weeks. A treatment cycle will consists of total of two doses per cycle. Part 2 of the study will enroll subjects with squamous cell type tumor to receive KHK2898 at a dose to be determined following completion of Part 1.

All subjects will receive study therapy until disease progression, the development of unacceptable toxicity, noncompliance or withdrawal of consent by the subject, or Investigator decision, up to a maximum of six cycles (approximately six months). After six cycles of KHK2898 therapy, the subject may continue to receive the drug after discussion with the Sponsor and determination that the subject is experiencing a best response of at least stable disease (SD) and is not experiencing any unacceptable toxicities or dose limiting toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a histopathological-documented, measurable or non-measurable, locally advanced unresectable primary or metastatic solid tumor unresponsive to standard therapy or for which there is no standard therapy available.
2. The subject has PD during or following the last treatment regimen as defined by the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1 guidelines)11.
3. The subject has a life expectancy >3 months.
4. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of ≤ 2 at study entry.
5. The subject is ≥ 18 years of age.
6. The subject has a pre-study echocardiogram or multigated acquisition scan with left ventricular ejection fraction ≥ 50%.
7. The subject has recovered to Grade ≤ 1 by the CTCAE v 4.0313, from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies for cancer, with the exception of alopecia or peripheral neuropathy (the latter of which must have resolved to Grade ≤ 2).
8. The subject has preserved organ function as defined below. All parameters must be evaluated within 7 days prior to the first dose of KHK2898.

   * 8-a) Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 ×Upper limits of normal (ULN), or ≤ 5.0 × ULN in subjects with metastatic liver disease
   * 8-b) Hemoglobin ≥ 9 g/dl (without transfusion in the preceding 7 days)
   * 8-c) Total bilirubin ≤ 1.5 × ULN
   * 8-d) Creatinine ≤ 1.5 × ULN
   * 8-e) ANC ≥ 1.5 × 109/L (unsupported by growth factors in the preceding 21 days)
   * 8-f) Platelets ≥ 100 × 109/L (without transfusion or growth factor in the preceding 7 days)
9. The subject has provided signed informed consent. Written informed consent must be obtained prior to performing any study-related procedures. For subject < 21 years old who is not married, written informed consent must be taken from the subject and his/her parents/ legal guardians.
10. Women of childbearing potential (WOCBP) must have a negative pregnancy test at study entry. Subjects not considered WOCBP are those without menses for 24 consecutive months, and those who have undergone hysterectomy and/or bilateral salpingo-oophorectomy. WOCBP must be willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study.

Exclusion Criteria:

1. The subject has received anti-cancer chemotherapy, hormonal therapy (other than LH-RH agonists/pure antagonists for prostate cancer, which are allowed to be continued if the subject has already been on one for at least 2 months at the time of enrollment), radiotherapy, immunotherapy, or investigational agents within 4 weeks (6 weeks for mitomycin C and nitrosoureas) prior to the first dose of KHK2898.
2. The subject has received monoclonal antibodies within 4 weeks of the first dose of KHK2898.
3. The subject had major surgery within 4 weeks prior to the first dose of KHK2898.
4. The subject has known symptomatic brain metastases (screening/baseline MRI of the brain is only required when there is clinical suspicion of central nervous system (CNS) involvement or past history of treated brain metastasis). Subjects with treated brain metastasis (radiotherapy and/or surgery) will be eligible if:

   * 4-a) They have completed treatment for their brain metastasis > 4 weeks prior to scheduled study treatment start date;
   * 4-b) They are neurologically stable;
   * 4-c) They are not receiving corticosteroids or corticosteroids in doses no greater than physiological replacement (e.g., dexamethasone < 1.5 mg/day); and
   * 4-d) They have a screening/baseline MRI scan of the brain that specifically verifies no evidence of CNS hemorrhage and no active gadolinium enhancing lesions; and
   * 4-e) Subjects with primary brain/CNS malignancy (e.g., gliomas, lymphomas) are excluded.
5. The subject has leptomeningeal disease.
6. The subject is pregnant (confirmed by beta human chorionic gonadotrophin [β-HCG]) or is lactating.
7. The subject has a significant uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring parenteral antibiotics, clinically significant cardiac disease [class II, III, or IV of the New York Heart Association classification (NYHA)],14 unstable angina pectoris, myocardial infarction within 6 months or is post angioplasty or stenting within 6 months, uncontrolled hypertension (i.e., systolic blood pressure (BP) > 150 mm Hg, diastolic BP > 90 mm Hg), found on two consecutive measurements separated by a 1-week period, clinically significant cardiac arrhythmia, or uncontrolled diabetes.
8. The subject has known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness.
9. The subject has known active hepatitis B or C or other active (non-malignant) liver disease.
10. The subject has a psychiatric illness, disability or social situation that would compromise the subject's safety, ability to provide consent, or limit his/her compliance with study requirements.
11. The subject has experienced a hypersensitivity reaction to monoclonal antibodies or other therapeutic proteins, and the reaction could not be controlled or prevented on subsequent infusion with standard therapies such as antihistamines, 5-HT3 antagonists, or corticosteroids.
12. The subject has a history of another primary cancer, with the exception of: a) curatively resected nonmelanomatous skin cancer, b) curatively treated cervical carcinoma in-situ, or c) other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 3 years.
13. The subject requires concomitant medication with any of the following prohibited medications: active prohibited anti neoplastic treatment other than the investigational product KHK2898; other anti-cancer therapies such as cytotoxic chemotherapy; anti-cancer hormonal therapy other than LH-RH agonists/pure antagonists for prostate cancer, which are allowed to be continued if the subject has already been on one for at least 2 months at the time of enrollment; immunotherapies including other monoclonal antibodies, interferons, cancer vaccines, etc; targeted small molecule anti-cancer therapies; and radiation therapy (radiation therapy should be completed prior to enrollment on this study).
14. Prior stem cell or bone marrow transplant.
15. Subjects received vaccination within 8 weeks from the first administration of KHK2898.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adverse Event collection and assessment | at least 28 days or up to 24 weeks
  Adverse Event collection and assessment will be done for all 54 potentially treated subjects to assess the safety, tolerability, and determine the DLTs, maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Evaluate preliminary evidence of efficacy | eight weeks
  Response and progression in subjects with solid tumors and measurable disease will be evaluated using RECIST criteria v 1.1. Evaluations will include: objective response (CR + PR) and clinical benefit (CR + PR + SD).
Profile of Pharmacokinetics | Pre-dose, 1, 2, 4, 6-8, 24, 48, 72, 96, 168, 240-288, 336 hours post-dose
  maximum concentration (Cmax), area under the curve (AUC), half-life (t1/2), clearance (Cl), and apparent volume of distribution in the terminal elimination phase (Vz).

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore, Singapore